CLINICAL TRIAL: NCT05497271
Title: Confirmation of Association Between Cystic Fluid Analysis With Pancreatic Cystic Lesions and Study of Its Application for Diagnosis, Treatment and Prognosis
Brief Title: Confirmation of Association Between Cystic Fluid Analysis With Pancreatic Cystic Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Other Study IDs: H-2206-213-1336
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Cyst; Molecular, Chemical Analysis of Cystic Fluid
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — cystic fluid DNA from cellular component in cystic fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through a comprehensive analysis of the pancreatic cystic fluid analysis, the role of the cystic fluid analysis is confirmed in terms of accurate diagnosis of pancreatic cysts, appropriate prediction of treatment response, and to select proper treatment indication through analytic results.

ELIGIBILITY:
Inclusion Criteria:

1. patients who diagnosed with pancreatic cystic lesion
2. patients who are able to acquire cystic fluid through EUS-FNA or surgery
3. patients aged 18 years and older

Exclusion Criteria:

1. patients who did not want to participate in this study
2. patients aged under 18 years old
3. severely mentally ill patients
4. pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were diagnosed with pancreatic cystic lesions and managed in Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy by cystic fluid analysis | up to 5 years after cystic fluid analysis
  diagnostic accuracy by cystic fluid analysis in comparison with pathologic diagnosis

SECONDARY OUTCOMES:
Overall survival | up to 5 years after cystic fluid analysis or surgical resection
  overall survival until death
Disease free survival | up to 5 years after cystic fluid analysis or surgical resection
  Period till tumor recurrence after surgical resection or intervention
Malignant transformation rate | up to 5 years after cystic fluid analysis
  the prevalence of malignant transformation during follow-up period (percent)
Prediction for treatment response in case of surgical resected or EUS-guided ethanol ablated pancreatic cysts | up to 5 years after cystic fluid analysis or EUS guided ablative therapy
  evaluation of treatment response for surgery of EUS guided therapy according to RECIST criteria v1.1
Cytology of cystic fluid | within 2 months after study enrollment
  result of cytology of cystic fluid
Chemical profile of CEA in cystic fluid | within 2 months after study enrollment
  level of CEA in cystic fluid
Chemical profile of Amylase in cystic fluid | within 2 months after study enrollment
  level of amylase in cystic fluid
Chemical profile of glucose in cystic fluid | within 2 months after study enrollment
  level of glucose in cystic fluid
DNA mutation profile of cystic fluid | within 2 months after study enrollment
  targeted NGS for KRAS, NRAS, CDKN2A, TP53, SMAD4, RNF43, PTEN, PIK3CA, VHL, Aneuploid

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea